CLINICAL TRIAL: NCT04548921
Title: Biomarker for Friedreich's Ataxia: An International, Multicenter, Observational, Longitudinal Protocol
Brief Title: Biomarker for Friedreich's Ataxia (BioFridA)
Acronym: BioFridA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BioFridA 06-2020
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: FXN Gene; FRDA; Hereditary Diseases
Keywords: Friedreich's Ataxia; Biomarker
MeSH Terms: conditions — Friedreich Ataxia; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Friedreich's Ataxia: Participant diagnosed with Friedreich's Ataxia aged between 2 and 50 years of age

SUMMARY:
International, multicenter, observational, longitudinal monitoring study to identify biomarker/s for Friedreich's Ataxia and to explore the clinical robustness, specificity, and long-term variability of these biomarker/s

DETAILED DESCRIPTION:
An ataxia is neurological disorder of balance and coordination resulting from dysfunctions of the cerebellum. Friedreich's ataxia (FRDA) is most common ataxia in white population, with an estimated prevalence of 2-4 cases per 100,000 individuals. With an average age of onset of 10-15 years, the disease is characterized by dysarthria, deep sensory loss, hypertrophic cardiomyopathy, spinocerebellar ataxia, pyramidal weakness, diabetes mellitus, and skeletal abnormalities.

FRDA is an autosomal recessive disorder caused by pathogenic variant/s in the FXN gene, which encodes the mitochondrial protein frataxin. In 98% of cases these are homozygous guanine-adenine-adenine (GAA) triplet repeat expansions in the ﬁrst intron of the FXN gene. The remaining cases are compound heterozygotes for a GAA repeat expansion plus a FXN point mutation or deletion. GAA repeat expansions suppress transcription of the FXN gene, leading to frataxin deﬁciency.

Until now there is no FDA-approved therapy for FRDA, but potential agents for treatment are in developing phases. As such, especially antioxidants like idebenone are tested in clinical trials as FRTA medication, whereas another study identified p38 inhibitors as potential therapeutic agents. Various clinical rating scales including the Scale for the Assessment and Rating of Ataxia (SARA), Friedreich's Ataxia Rating Scale (FARS), and the International Cooperative Ataxia Rating Scale (ICARS) have been used as trial endpoints in FRDA, but these measurements have limited sensitivity to disease progression over 12 months. Furthermore, there are no validated, objective central or peripheral nervous system biomarkers of disease progression for use in clinical trials as intermediate endpoints.

It is the goal of the BioFridA study to identify, validate, and monitor FRDA biomarker/s.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant or parent/ legal guardian
* The participant is aged between 2 and 50 years of age
* The diagnosis of Friedreich's Ataxia (FRDA) is genetically confirmed by CENTOGENE

Exclusion Criteria:

* Informed consent is not obtained from the participant and parent/ legal guardian
* The participant is younger than 2 years or older than 50 years of age
* The diagnosis of FRDA is not genetically confirmed by CENTOGENE

Ages: 2 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with Friedreich's Ataxia
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of Friedreich's Ataxia biomarker/s | 36 months
  All samples will be analyzed for the identification of potential biomarkers via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s.

SECONDARY OUTCOMES:
Exploring the clinical robustness, specificity, and long-term variability of Friedreich's Ataxia biomarker/s | 36 months
  All samples will be analyzed for the identification of potential biomarkers via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof. Dr., Study Chair — CENTOGENE GmbH
Locations (1):
- American University of Science and Technology, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided